CLINICAL TRIAL: NCT04577820
Title: Evaluation of Efficacy and Safety of Garetosmab in Japanese Adult Patients With Fibrodysplasia Ossificans Progressiva
Brief Title: Study to Assess the Efficacy and Safety of Garetosmab in Japanese Adult Patients With Fibrodysplasia Ossificans Progressiva (FOP)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Phase 2 Study R2477-FOP-1940 has been withdrawn and the next phase of the development program is being planned
Sponsor: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R2477-FOP-1940
Record Dates: First submitted 2020-09-30; First posted 2020-10-08 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Fibrodyplasia Ossificans Progressiva (FOP); Heterotopic Ossification (HO)
MeSH Terms: conditions — Ossification, Heterotopic

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- garetosmab (Experimental)
  Interventions: Drug: garetosmab

INTERVENTIONS:
Drug: garetosmab — Repeated doses administered intravenously (IV) every four weeks (Q4W)
  Other Names: REGN2477

SUMMARY:
The primary safety objective of the study is to assess the safety and tolerability of garetosmab in Japanese male and female adult patients with FOP.

The primary efficacy objective of the study is to assess the effect of garetosmab on Heterotopic ossification (HO) in Japanese adult patients with FOP, as determined by the number of new heterotopic bone lesions identified by computed tomography (CT).

ELIGIBILITY:
Key Inclusion Criteria:

* Clinical diagnosis of FOP (based on findings of congenital malformation of the great toes, episodic soft tissue swelling, and/or progressive HO)
* Confirmation of FOP diagnosis with documentation of any Type I activin A receptor (ACVR1) mutation
* FOP disease activity, as defined in the protocol, within 1 year of screening visit
* Willing and able to undergo PET and CT imaging procedures and other procedures as defined in this study
* Able to understand and complete study-related questionnaires and diaries (assistance from caregivers is allowed)

Key Exclusion Criteria:

* Patient has significant concomitant illness or history of significant illness such as but not limited to cardiac, renal, rheumatologic, neurologic, psychiatric, endocrine, metabolic, or lymphatic disease, that in the opinion of the study investigator might confound the results of the study or pose additional risk to the patient by their participation in the study
* Previous history or diagnosis of cancer
* Severely impaired renal function defined as estimated glomerular filtration rate <30 mL/min/1.73 m2 calculated by the Modification of Diet in Renal Disease equation (1 retest is allowed)
* Uncontrolled diabetes defined as hemoglobin A1C (HbA1c) >9% at screening (1 retest allowed)
* History of severe respiratory compromise, as defined in protocol
* Concurrent participation in another interventional clinical study or a non-interventional study with radiographic measures or invasive procedures
* Pregnant or breastfeeding women

NOTE: Other protocol defined inclusion/exclusion criteria apply.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-13 (Estimated); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-10-08 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse event (TEAEs) | Through week 28
Number of new HO lesions as assessed by CT | At week 28

SECONDARY OUTCOMES:
Total volume of new HO lesions as assessed by CT | At week 28
Number of new HO lesions as assessed by positron emission tomography (PET) | At week 28
Total lesion activity in new HO lesions as assessed by PET | At week 28
Percent of patients with new HO lesions as assessed by CT | At week 28
Percent of patients with new HO lesions as assessed by PET | At week 28
Percent of patients with investigator-assessed flare-ups | Baseline to week 28
Percent of patients with investigator-assessed flare-ups | Baseline to week 56
Percent of patients with flare-ups assessed by patient e-diary | Baseline to week 28
Percent of patients with flare-ups assessed by patient e-diary | Baseline to week 56
Number of new HO lesions as assessed by CT | At week 56
Total volume of new HO lesions as assessed by CT | At week 56
Percent of patients with new HO lesions as assessed by CT | At week 56
Number of new HO lesions as assessed by PET | At week 56
Total lesion activity in new HO lesions as assessed by PET | At week 56
Percent of patients with new HO lesions as assessed by PET | At week 56
Change in mean maximum standard uptake volume (SUVmax) of individual active HO site(s) by PET | Baseline and week 28
Change in mean maximum standard uptake volume (SUVmax) of individual active HO site(s) by PET | Baseline and week 56
Percent change in mean maximum standard uptake volume (SUVmax) of individual active HO site(s) by PET | Baseline and week 28
Percent change in mean maximum standard uptake volume (SUVmax) of individual active HO site(s) by PET | Baseline and week 56
Change in total lesion activity by PET | Baseline and week 28
Change in total lesion activity by PET | Baseline and week 56
Percent change in total lesion activity by PET | Baseline and week 28
Percent change in total lesion activity by PET | Baseline and week 56
Change in the total volume of HO lesions as assessed by CT | Baseline and week 28
Change in the total volume of HO lesions as assessed by CT | Baseline and week 56
Percent change in the total volume of HO lesions as assessed by CT | Baseline and week 28
Percent change in the total volume of HO lesions as assessed by CT | Baseline and week 56
Change in number of HO lesions as assessed by PET | Baseline and week 28
  HO lesions defined as target and new lesions relative to baseline.
Change in number of HO lesions as assessed by PET | Baseline and week 56
  Defined above
Change in the number of HO lesions detectable by CT | Baseline and week 28
  Defined above
Change in the number of HO lesions detectable by CT | Baseline and week 56
  Defined above
Time-weighted average (standardized area under curve [AUC]) change in daily pain due to FOP, as measured using the daily numeric rating scale (NRS) | Baseline through week 28
  The NRS is a categorical rating scale used by patients to rate their pain associated with FOP. Patients will be asked to rate their pain on a scale that ranges from "0" (no pain) to "10" (worst possible pain).
Time-weighted average (standardized AUC) change in daily pain due to FOP, as measured using the daily NRS | Baseline through week 56
Total dosage of glucocorticoids use | Through week 56
Incidence and severity of TEAEs | Through week 56
Concentration of total activin A in serum over time | Through week 56
Pharmacokinetic (Pk) Profile - concentrations of garetosmab in serum over time | Through week 56
Immunogenicity as measured by Anti-drug antibodies (ADA) to garetosmab over time | Through week 28
Percent change from baseline in biomarkers of bone formation levels in serum | Through week 28

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial Management, Study Director — Regeneron Pharmaceuticals

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie publicly available results will be considered for sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: When Regeneron has received marketing authorization from major health authorities (e.g., FDA, European Medicines Agency (EMA), Pharmaceuticals and Medical Devices Agency (PMDA), etc.) for the product and indication, has made the study results publicly available (e.g., scientific publication, scientific conference, clinical trial registry), has the legal authority to share the data, and has ensured the ability to protect participant privacy.
Access Criteria: Qualified researchers can submit a proposal for access to individual patient or aggregate level data from a Regeneron-sponsored clinical trial through Vivli. Regeneron's Independent Research Request Evaluation Criteria can be found at: https://www.regeneron.com/sites/default/files/Regeneron-External-Data-Sharing-Policy-and-Independent-Research-Request-Evaluation-Criteria.pdf
URL: https://vivli.org/